CLINICAL TRIAL: NCT00288002
Title: A Randomized Phase III Study Exploring the Efficacy of Capecitabine Given Concomitantly or in Sequence to EC-Doc With or Without Trastuzumab as Neoadjuvant Treatment of Primary Breast Cancer
Brief Title: Combination Chemotherapy With or Without Capecitabine and/or Trastuzumab Before Surgery in Treating Women With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455125; GBG-GEPARQUATTRO; GBG-40; EU-205101; AVENTIS-GBG-GEPARQUATTRO; ROCHE-AVENTIS-GBG-GEPARQUATTRO; EUDRACT-2005-001546-17
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IA breast cancer; stage IB breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; HER2-negative breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Trastuzumab; Capecitabine; Cyclophosphamide; Docetaxel; Epirubicin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Biological: trastuzumab
Drug: capecitabine
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, cyclophosphamide, docetaxel, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Giving combination chemotherapy together with monoclonal antibodies before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving monoclonal antibodies after surgery may kill any tumor cells that remain after surgery. It is not yet known whether combination chemotherapy is more effective with or without capecitabine and/or trastuzumab in treating breast cancer.

PURPOSE: This randomized phase III trial is studying epirubicin, cyclophosphamide, and docetaxel to compare how well they work with or without capecitabine and/or trastuzumab before surgery in treating women with stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the pathologic complete response rates in women with stage I-III primary breast cancer treated with neoadjuvant epirubicin hydrochloride, cyclophosphamide, and docetaxel with versus without capecitabine followed by surgery .
* Compare the pathologic complete response rates in women with HER-2/neu-positive tumors receiving trastuzumab (Herceptin®) simultaneously with neoadjuvant epirubicin hydrochloride, cyclophosphamide, and docetaxel to women with HER-2/neu-negative tumors receiving neoadjuvant chemotherapy only.

Secondary

* Determine the toxicity of these regimens in these patients.
* Determine the disease-free (loco-regional and distant) survival and overall survival of patients treated with these regimens.
* Determine the disease-free (loco-regional and distant) survival and overall survival of patients treated with or without trastuzumab.
* Determine the breast conservation rate in patients treated with these regimens.
* Determine the frequency of the use of sentinel node biopsy for selecting patients for neoadjuvant chemotherapy.
* Compare the frequency of sentinel node biopsies at surgery after neoadjuvant chemotherapy in each arm.
* Determine the pathologic complete response rates to each regimen in the subgroup of patients with locally advanced (T4a-d, N0-3, M0) breast cancer.
* Determine the response rate (complete response, partial response, or no change) at surgery (by imaging methods and by histopathological exam) in patient subgroups according to their response after four treatments with epirubicin hydrochloride and cyclophosphamide.
* Determine the intention for the use of neoadjuvant chemotherapy, in terms of freedom from disease, avoiding mastectomy, improving breast conservation, and gaining information about efficacy.

OUTLINE: This is a randomized, controlled, open-label, multicenter study. Patients are stratified according to participating site, clinical response after 4 courses of epirubicin hydrochloride and cyclophosphamide (complete response vs partial response vs no change), HER-2/neu-status (negative vs 3+ by immunohistochemistry [IHC] or positive by fluorescence in situ hybridization [FISH]), estrogen receptor (ER)/progesterone receptor (PR) status (ER or PR positive vs ER and PR negative), and extent of disease (T4 or N3 vs T1-3 and N0-2).

All patients receive epirubicin hydrochloride IV over 30-60 minutes and cyclophosphamide IV over 60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are then randomized to 1 of 3 treatment arms.

* Arm I: Patients receive docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive docetaxel as in arm I. Patients also receive oral capecitabine twice daily on days 1-14. Treatment with docetaxel and capecitabine repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive docetaxel as in arm I. Patients then receive oral capecitabine twice daily on days 1-14. Treatment with capecitabine repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with HER-2/neu-positive tumors also receive trastuzumab (Herceptin®) IV over 90 minutes on day 1 of each course of chemotherapy (during treatment with epirubicin hydrochloride and cyclophosphamide AND during randomized treatment).

Within 2 weeks after completion of chemotherapy, all patients undergo surgery. Within 2 weeks after surgery, patients with HER-2/neu-positive tumors resume trastuzumab treatment for up to 1 year.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 1,500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unilateral or bilateral primary breast cancer

  * Meets 1 of the following staging criteria:

    * Clinical stage T4 or T3 disease
    * Clinical stage T1 and pathologic stage N+ by sentinel lymph node biopsy OR clinical stage T2, N+ disease AND estrogen receptor (ER) or progesterone receptor (PR) positive tumor
    * ER and PR negative tumor (T1-4, N0-3, M0)
* Disease confirmed by core biopsy

  * No fine-needle aspiration or incisional biopsy
* Bidimensionally measurable disease*

  * Tumor lesion palpable and measures ≥ 2 cm OR tumor lesion ≥ 1 cm in maximum diameter by sonography

    * For inflammatory disease, extent of inflammation can be used as measurable lesion NOTE: *In patients with multifocal or multicentric breast cancer, the largest lesion should be measured
* Candidate for adjuvant chemotherapy

  * No low- or moderate-risk patients who are doubtful candidates for adjuvant chemotherapy and do not fulfill the staging criteria
* Known HER-2/neu status by core biopsy

  * HER-2/neu positive tumor is defined as +3 by immunohistochemistry [IHC] OR positive by fluorescence in situ hybridization (FISH)
* No evidence of distant metastasis
* Hormone receptor status:

  * ER- or PR-positive tumor OR ER- and PR-negative tumor

PATIENT CHARACTERISTICS:

* No male patients
* Menopausal status not specified
* Karnofsky performance status 80-100%
* Life expectancy ≥ 10 years (disregarding diagnosis of cancer)
* Normal cardiac function confirmed by ECG
* LVEF ≥ 55% by cardiac ultrasound
* Neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase (AP) ≤ 5 times ULN OR
* AP ≤ 2.5 times ULN AND AST and/or ALT ≤ 1.5 times ULN
* Creatinine ≤ 2 mg/dL
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No motor or sensory neuropathy ≥ grade 2
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* No New York Heart Association class II-IV congestive heart failure
* No coronary artery disease
* No history of myocardial infarction
* No uncontrolled arterial hypertension (i.e., blood pressure ≥ 160/90 mm Hg despite antihypertensive therapy)
* No rhythm abnormalities requiring permanent therapy
* No history of significant neurological or psychiatric disorders including psychotic disorders, dementia, or seizures that would preclude giving informed consent
* No active infection
* No active peptic ulcer
* No unstable diabetes mellitus or insulin-dependent type II diabetes mellitus
* No other serious illness or medical condition
* No known hypersensitivity reaction to investigational compounds or incorporated substances
* No definite contraindications for the use of corticosteroids
* No known dihydropyrimidine dehydrogenase deficiency
* Must be fit for anthracycline/taxane-containing chemotherapy

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for any malignancy
* No prior radiation therapy for breast cancer
* No concurrent bisphosphonates during chemotherapy

  * Bisphosphonates allowed postoperatively
* No chronic treatment with corticosteroids unless it is initiated > 6 months prior to study entry and is given at low doses (≤ 20 mg methylprednisolone or equivalent)
* No concurrent amifostine during chemotherapy
* No concurrent cardioprotectors (e.g., dexrazoxane) during chemotherapy
* No concurrent sex hormone therapy
* No concurrent virostatic agents (e.g., sorivudine or brivudine)
* No concurrent aminoglycosides
* No other concurrent experimental drugs or anticancer therapy
* At least 30 days since prior participation in another clinical trial with any investigational (not marketed) drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2005-01

PRIMARY OUTCOMES:
Pathologic complete response

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, MD, Principal Investigator — GBG Forschungs GmbH
Locations (1):
- Universitaetsfrauenklinik Frankfurt, Neu-Isenburg, Germany

REFERENCES:
- [Result] Untch M, Rezai M, Loibl S, Fasching PA, Huober J, Tesch H, Bauerfeind I, Hilfrich J, Eidtmann H, Gerber B, Hanusch C, Kuhn T, du Bois A, Blohmer JU, Thomssen C, Dan Costa S, Jackisch C, Kaufmann M, Mehta K, von Minckwitz G. Neoadjuvant treatment with trastuzumab in HER2-positive breast cancer: results from the GeparQuattro study. J Clin Oncol. 2010 Apr 20;28(12):2024-31. doi: 10.1200/JCO.2009.23.8451. Epub 2010 Mar 22. PMID 20308670
- [Result] von Minckwitz G, Rezai M, Loibl S, Fasching PA, Huober J, Tesch H, Bauerfeind I, Hilfrich J, Eidtmann H, Gerber B, Hanusch C, Kuhn T, du Bois A, Blohmer JU, Thomssen C, Dan Costa S, Jackisch C, Kaufmann M, Mehta K, Untch M. Capecitabine in addition to anthracycline- and taxane-based neoadjuvant treatment in patients with primary breast cancer: phase III GeparQuattro study. J Clin Oncol. 2010 Apr 20;28(12):2015-23. doi: 10.1200/JCO.2009.23.8303. Epub 2010 Mar 22. PMID 20308671
- [Result] Witzel I, Loibl S, von Minckwitz G, Mundhenke C, Huober J, Hanusch C, Henschen S, Hauschild M, Lantzsch T, Tesch H, Latos K, Just M, Hilfrich J, Barinoff J, Eulenburg CZ, Roller M, Untch M, Muller V. Monitoring serum HER2 levels during neoadjuvant trastuzumab treatment within the GeparQuattro trial. Breast Cancer Res Treat. 2010 Sep;123(2):437-45. doi: 10.1007/s10549-010-1030-9. Epub 2010 Jul 10. PMID 20623180
- [Result] Riethdorf S, Loibl S, Komor M, et al.: Incidence and kinetics of circulating tumor cells in breast cancer patients treated with primary systemic therapy including trastuzumab for patients with HER2-positive tumors a translational project within the study GeparQuattro. [Abstract] Breast Cancer Res Treat 106 (1): A-5025, S214, 2007.
- [Result] von Minckwitz G, Rezai M, Loibl S, et al.: Evaluating the efficacy of capecitabine given concomitantly or in sequence to epirubicin/cyclophosphamide docetaxel as neoadjuvant treatment for primary breast cancer. First efficacy analysis of the GBG/AGO intergroup-study GeparQuattro. [Abstract] Breast Cancer Res Treat 106 (1): A-79, S21-2, 2007.
- [Derived] von Minckwitz G, Rezai M, Fasching PA, Huober J, Tesch H, Bauerfeind I, Hilfrich J, Eidtmann H, Gerber B, Hanusch C, Blohmer JU, Costa SD, Jackisch C, Paepke S, Schneeweiss A, Kummel S, Denkert C, Mehta K, Loibl S, Untch M. Survival after adding capecitabine and trastuzumab to neoadjuvant anthracycline-taxane-based chemotherapy for primary breast cancer (GBG 40--GeparQuattro). Ann Oncol. 2014 Jan;25(1):81-9. doi: 10.1093/annonc/mdt410. Epub 2013 Nov 21. PMID 24273046
- [Derived] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812